## **MELT-HF NCT02620384**

MEtolazone as Early add on Therapy for acute decompensated Heart Failure.

A single center pilot study.

Muhammad A. Chaudhry, MD

## STATISTICAL ANALYSIS (UPDATED 12/4/2018) Statistical Methods

- Power Analysis: In the DOSE trial urine output at 72 hours was 4200ml with a standard deviation of 3200 ml.
- With 1:1 randomization, there is a power of more than 80% to detect a difference of 3000-4000 ml between the groups at 48 hours and at least 200 patients will be enrolled to achieve statistical significance.
- The demographics to the two groups were compared with Student's T test for continuous variables and Chi Square for categorical variables. There were no significant differences in age, gender, race or NYHA enrollment.
- ■Primary and secondary outcomes were compared with Student's T tests and Repeated Measures ANOVA (for longitudinal data) with between subjects variable.